CLINICAL TRIAL: NCT02766816
Title: A Phase III, Observer Blind, Active Controlled, Randomized, Clinical Study Comparing Safety and Immunogenicity of BBio Bivalent Oral Polio Vaccine With a Licensed Bivalent Oral Polio Vaccine
Brief Title: A Clinical Study Comparing Safety and Immunogenicity of bOPV of Bilthoven Biologicals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bilthoven Biologicals (Industry)
Collaborators: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OPV-03/PR-15106; PR-15106 (Other: icddr,b)
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Immune Response to Oral Polio Vaccine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1 Study - BBio bOPV (Experimental)
  Interventions: Biological: Part 1 study - BBio bOPV
- Part 1 Study - Licensed bOPV (Active Comparator)
  Interventions: Biological: Part 1 study - Licensed bOPV
- Part 2 Study - BBio bOPV Lot 1 (Experimental)
  Interventions: Biological: Part 2 study - BBio bOPV Lot 1
- Part 2 Study - BBio bOPV Lot 2 (Experimental)
  Interventions: Biological: Part 2 study - BBio bOPV Lot 2
- Part 2 Study - BBio bOPV Lot 3 (Experimental)
  Interventions: Biological: Part 2 study - BBio bOPV Lot 3
- Part 2 Study - Licensed bOPV (Active Comparator)
  Interventions: Biological: Part 2 study - Licensed bOPV

INTERVENTIONS:
Biological: Part 1 study - BBio bOPV — A single dose of 2 drops (0.1 ml) orally of BBio bOPV to 20 children 60 to 83 months of age.
  Arms: Part 1 Study - BBio bOPV
Biological: Part 2 study - BBio bOPV Lot 1 — Three doses of 2 drops (0.1 ml) orally of BBio bOPV Lot 1 to 270 infants at 6-8, 10-12 and 14-16 weeks of age.
  Arms: Part 2 Study - BBio bOPV Lot 1
Biological: Part 2 study - BBio bOPV Lot 2 — Three doses of 2 drops (0.1 ml) orally of BBio bOPV Lot 2 to 270 infants at 6-8, 10-12 and 14-16 weeks of age.
  Arms: Part 2 Study - BBio bOPV Lot 2
Biological: Part 2 study - BBio bOPV Lot 3 — Three doses of 2 drops (0.1 ml) orally of BBio bOPV Lot 3 to 270 infants at 6-8, 10-12 and 14-16 weeks of age.
  Arms: Part 2 Study - BBio bOPV Lot 3
Biological: Part 2 study - Licensed bOPV — Three doses of 2 drops (0.1 ml) orally of a licensed bOPV to 270 infants at 6-8, 10-12 and 14-16 weeks of age.
  Arms: Part 2 Study - Licensed bOPV
Biological: Part 1 study - Licensed bOPV — A single dose of 2 drops (0.1 ml) orally of a licensed bOPV to 20 children 60 to 83 months of age.
  Arms: Part 1 Study - Licensed bOPV

SUMMARY:
Bilthoven Biologicals has developed a new bivalent oral polio vaccine (bOPV) containing World Health Organization (WHO) approved Sabin strains of poliovirus type 1 and type 3. This study will assess non-inferiority of bOPV manufactured by BBio to that of licensed bOPV. This study will also assess lot-to-lot consistency among three lots of BBio bOPV.

DETAILED DESCRIPTION:
Bilthoven Biologicals has developed a new bivalent OPV containing WHO approved Sabin strains of poliovirus type 1 and type 3. This phase III study will be conducted in two parts:

Part 1 - 40 children of 60 to 83 months of age will be given single dose of BBio bOPV or licensed bOPV in 1:1 ratio. Primary objective is to assess safety of BBio bOPV.

Part 2 - A total of 1080 infants of 42 to 56 days of age will be randomized to receive three doses of either BBio bOPV from one of the three lots or a licensed bOPV in 1:1:1:1 ratio as primary immunization series at 6, 10 and 14 weeks of age.

Primary objective of this study is to assess non-inferiority of bOPV manufactured by BBio to that of licensed bOPV in terms of seroconversion. This study also will assess lot-to-lot consistency among three lots of BBio bOPV.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy children of both sexes of age 5 to 6 years (60-83 months) at the time of vaccination and who have received at least 3 doses of trivalent oral polio vaccine (tOPV) based upon documentation (Study Part 1).
2. Normal healthy infants of both sexes of age 6-8 weeks (42-56 days) at the time of the first vaccination and have not received oral polio vaccine (OPV) previously based upon documentation (Study Part 2).
3. Parents/legal guardians of participants willing to give written informed consent and willing to comply with study protocol.
4. Free of obvious health problems as established by medical history and screening evaluation including clinical examination.
5. Resident of study area.

Exclusion Criteria:

1. Participation in another clinical trial in the 4 weeks preceding the (first) trial vaccination or planned participation in another clinical trial during the present trial period.
2. A diagnosis or suspicion of congenital or acquired immunodeficiency disorder, malignancy, receiving immunosuppressive therapy such as systemic corticosteroids therapy for a period of ≥ 1 week either in the participant or in an immediate family member.
3. A diagnosis or suspicion of bleeding disorder that would contraindicate collection of blood by venipuncture.
4. Acute or persistent diarrhea (defined as diarrhea that lasts 14 days or longer), infection or illness at the time of enrollment (6-8 weeks of age) that would require participant's admission to a hospital or would contraindicate provision of OPV.
5. Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit.
6. Infants from multiple births (i.e. twins).
7. History of allergy or systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the study vaccines or a vaccine containing the same substances.
8. Chronic illness at a stage that could interfere with trial conduct or completion.
9. Planned administration/ administration of a vaccine not foreseen by the study protocol during the study period with the exception of routine Expanded Program on Immunization (EPI) program vaccines including pneumococcal vaccine, and rotavirus vaccine (Polio vaccines are not allowed during the study period).
10. Blood or blood-derived products received in the past.
11. Any vaccination one week preceding the trial vaccination.
12. Presence of significant malnutrition (< -3 standard deviation [SD] weight for length) or acute or chronic, clinically significant pulmonary, endocrine, autoimmune, cardiovascular, metabolic, hepatic or renal functional abnormality, as determined by medical history, and physical examination, which in the opinion of the investigator, might interfere with the study objectives
13. History of any neurological disorder or history of seizure (febrile or afebrile), or encephalopathy, encephalitis, hypotonic-hyporesponsive episode.
14. Febrile illness or acute illness on the day of inclusion is temporary exclusion criterion.
15. Participant with any other condition, which, in the opinion of the investigator would jeopardize the safety or rights of the participant participating in the study or making it unlikely the participant, could complete the protocol.

Ages: 42 Days to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1120 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Part 1 study: Frequency of adverse events (AEs) | 4 Days
  Safety of single dose of BBio bOPV will be assessed at 4 days after vaccination.
Part 2 study: Percentage of seroconversion to poliovirus type 1 and type 3 | one month after dose 3
  Percentage of seroconversion to poliovirus type 1 and type 3 one month after administration of third dose of the BBio bOPV to that of control group bOPV to assess non-inferiority of BBio bOPV to that of a licensed bOPV.
Part 1 study: Frequency of AEs and serious AEs (SAEs) | 28 days
  Safety of single dose of BBio bOPV will be assessed at 28 days after vaccination.

SECONDARY OUTCOMES:
Part 1 study: Percentage of seroprotection to poliovirus type 1 and type 3 | one month
  Percentage of seroprotection to poliovirus type 1 and type 3 one month after administration of single dose of the BBio bOPV to that of control group.
Part 1 study: Geometric mean titers (GMTs) of poliovirus neutralizing antibody (PVNA) to poliovirus type 1 and type 3 | one month
  GMTs of PVNA to poliovirus type 1 and type 3 at one month after administration of single dose of the BBio bOPV.
Part 2 study: GMTs of serum PVNA for the three lots of BBio bOPV | one month after dose 3
  Serum PVNA concentrations expressed as GMTs for the BBio bOPV to assess equivalence in manufacturing consistency among three current Good Manufacturing Practices (cGMP) lots of the BBio bOPV.
Part 2 study: GMTs of PVNA to poliovirus type 1 and type 3 | one month after dose 3
  Comparison of GMTs of PVNA to poliovirus type 1 and type 3 at one month after administration of third dose of the BBio bOPV to that of control group bOPV.
Part 2 study: Percentage of seroprotection to poliovirus type 1 and type 3 | one month after dose 3
  Percentage of seroprotection to poliovirus type 1 and type 3 one month after administration of third dose of the BBio bOPV to that of control group bOPV.
Part 2 study: Frequency of adverse events within 4 days following the administration of each dose of vaccine | 4 days after each dose of vaccine
  Frequency of adverse events within 4 days following the administration of each dose of vaccine
Part 2 study: Frequency of adverse events and serious adverse events | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, MBBS, MPH, Principal Investigator — International Center for Diarrheal Disease Research
Locations (1):
- Matlab Hospital Research Centre, International Center for Diarrheal Disease Research, Matlab, Matlab South, Chandpur District, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaman K, Kingma R, Yunus M, van Straaten I, Mekkes D, Bouwstra X, Gunale B, Kulkarni PS. Safety, immunogenicity and lot-to-lot consistency of a new Bivalent Oral Polio Vaccine (bOPV) in healthy Infants: Results of a Phase III, observer blind, randomized, controlled clinical study. Vaccine. 2019 Jul 18;37(31):4275-4280. doi: 10.1016/j.vaccine.2019.06.048. Epub 2019 Jun 22. PMID 31235374